CLINICAL TRIAL: NCT04057924
Title: Therapeutic Abstention and Surveillance of Intra-epithelial Histological Lesions of High Grade Cervical CIN2 (Cervical Intraepithelial Neoplasia Grade 2). SUIVICIN
Acronym: SUIVICIN
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/03
Record Dates: First submitted 2019-07-04; First posted 2019-08-15 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: HPV Infection; Cervical Cancer
Keywords: HPV; alternative to surgery; cervical cancer
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CIN 2 women: Non-interventional monocentric prospective study taking place at the Bordeaux University Hospital where women with a CIN2 meeting the eligibility criteria will benefit from abstention from treatment and surveillance for at least 2 years
  Interventions: Other: abstention from CIN2 treatment and surveillance for at least 2 years

INTERVENTIONS:
Other: abstention from CIN2 treatment and surveillance for at least 2 years — Non-interventional monocentric prospective study taking place at the Bordeaux University Hospital where women with a CIN2 meeting the eligibility criteria will benefit from abstention from treatment and surveillance for at least 2 years

SUMMARY:
This study proposes to describe and evaluate the rate of spontaneous regression of CIN2 at 2 year of follow up in women between 18 and 39 year old. This follow-up is proposed as an alternative to the treatment of reference (conization) with a possible extension to 4 years

DETAILED DESCRIPTION:
The INCa recommendations of December 2016 propose the destruction or abstention-monitoring of high-grade histological cervical lesions (HSIL) as an alternative to conization under certain conditions. These are women under 30 years old, with a small lesion in colposcopy, without any sign of invasion, with a squamocolumnar junction seen. These women must accept the principle of regular monitoring by cytology and colposcopy +/- biopsy every 6 months for a maximum of 2 years. HSIL group 2 histological entities CIN2 and CIN3. It is recognized that CIN2 are associated with CIN1 and CIN3 biology whose diagnosis is the result of the subjectivity of colposcopy allowing cervical biopsy and the variability of pathological interpretation due to poor reproducibility of histological diagnosis. CIN2 regress spontaneously in more than 50% of cases at 1 year, either completely (no lesion) or partially (LSIL low grade lesions). No invasive lesions are diagnosed over 2-year observation periods. Among the clinical, pathological and virological criteria, only the initial HPV genotyping seems to have a prognostic influence. There is therefore no strong scientific argument for routine conization in a woman over 30 years of age with a CIN2 lesion extended over more than two quadrants. In addition, conization is associated with an obstetrical risk (prematurity) and post-therapeutic colposcopic cervical stenosis complicates subsequent monitoring in case of abnormal smears. These considerations encourage the extension of the indications of abstention monitoring in the management of women with CIN2 wishing to procreate with an extension of the age to 39 year old, with no limit of size of the lesion and to satisfactory colposcopy

ELIGIBILITY:
Inclusion Criteria:

* CIN2 confirmed by biopsy, age between 18 and 39 years,
* satisfactory colposcopy identifying the junction and the lesion,
* affiliated person or beneficiary of a social security scheme,
* having given their oral agreement and authorization to the processing of their data.

Exclusion Criteria:

* Pregnancy in progress,
* history of conization,
* atypical or atypical glandular cells or cancer incidentally discovered during smear,
* prophylactic vaccination against HPV,
* active systemic infection requiring treatment, history of HIV infection, congenital or acquired immunodepression,
* long-term treatment with corticosteroids or immunosuppressants, placement under safeguard of justice,
* non-compliance with protocol requirements, in particular a supposed lack of compliance with long-term follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with a CIN2 meeting the eligibility criteria will benefit from abstention from treatment and surveillance for at least 2 years
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-08-23 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
rate of spontaneous regression of CIN2 at 2 years | 2 years
  Rate of spontaneous regression of CIN2 at 2 years, either complete (disappearance of the lesion) or partial (<lesions of low grade LSIL).

SECONDARY OUTCOMES:
rate of regression of CIN2 at 4 years | 4 years
  rate of regression of CIN2 at 4 years in women who responded to the main rate of regression of CIN2 at 4 years in women who responded to the main objective (disappearance of the lesion or lesions <low grade LSIL) and monitored for 2 more years
4-year regression rate of CIN2 that persisted for 2 years | 1, 2, 3 and 4 years
  evaluate the 4-year regression rate of CIN2 that persisted for 2 years in women who had not been treated with conization
HPV viral expression | 1, 2, 3 and 4 years
  Binary criteria: yes / No

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No